CLINICAL TRIAL: NCT06141525
Title: Safety and Efficacy of Remote Ischemic Conditioning for Patients Taking Off-pump Coronary Artery Bypass Grafting (IMPROVE): A National, Multi-center, Randomized, Controlled, Open-label, Blinded-endpoint Trial
Brief Title: Safety and Efficacy of Remote Ischemic Conditioning for Patients Taking Off-pump Coronary Artery Bypass Grafting
Acronym: IMPROVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Beijing Anzhen Hospital (Other); People's Hospital of Qinghai Province (Unknown); The Second Hospital of Yulin City (Unknown); Baoji Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: XJTU1AF2022LSK-427-01
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Bypass Grafting; Remote Ischemic Conditioning; Ischemia-Reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Experimental): In the RIC group, patients will undergo RIC training in the 3 days before and 7 days after the CABG surgery.
  Interventions: Device: Remote ischemic conditioning
- Control group (No Intervention): In the control group, a blood pressure cuff, same as the cuff in the RIC group, will be placed on both upper arms of the patients but only pressurized to 60 mmHg. The rest of the procedures will be the same.

INTERVENTIONS:
Device: Remote ischemic conditioning — An automatic programmed blood pressure cuffs will be placed on two upper limbs of the patient and pressurized to 200 mmHg (or at least 20 mmHg higher than the systolic blood pressure if the systolic blood pressure of the patient is above 180 mmHg) with 5 minutes of pressurization and 5 minutes of rest. One pressurization with rest is deemed as one cycle (10 minutes), and 4 cycles will be performed each time (for a total of 40 minutes).
  Arms: RIC group

SUMMARY:
Remote ischemic conditioning (RIC) is the process of repeated ischemia and reperfusion in the peripheral vessels, which is proved in reducing IRI in vital organs. This IMPROVE trial plans to enroll 648 patients who are diagnosed with coronary artery disease and are going to take off-pump CABG in five centers in China, to access whether RIC can and improve short-term prognosis.

DETAILED DESCRIPTION:
Remote ischemic conditioning (RIC) is the process of repeated ischemia and reperfusion in the peripheral vessels, which is proved in reducing IRI in vital organs. However, the effect of RIC in patients undergoing off-pump CABG is still unclear. This IMPROVE trial plans to enroll 648 patients who are diagnosed with coronary artery disease and are going to take off-pump CABG in five centers in China, to access whether RIC can and improve short-term prognosis. Patients will be randomly assigned into RIC group and control group. The primary outcome is the occurrence of the major adverse cardiovascular and cerebrovascular events (MACCE) within the 3-month follow-up. The MACCE is defined as all-cause of death, myocardial infarction, stroke and coronary revascularization surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with coronary artery disease and require off-pump CABG surgery.
* Between 18 and 75 years old;
* Normal left ventricular systolic function (ejection fraction >40%) and left ventricular end-diastolic internal diameter (<60 mm) in the cardiac ultrasound tests;
* No or mild heart valve and great vessel abnormalities which do not require surgical intervention;
* Participants or their authorized relatives agree to participate in the clinical trial and sign the informed consent.

Exclusion Criteria:

* Severe tissue injuries.
* Myalgia, fractures and other peripheral vascular lesions.
* Bypass graft being the radial artery.
* Stenosis or severe malformations of the subclavian, jugular and femoral arteries and veins.
* Previous vagus nerve trunk dissection or vagus nerve block surgery.
* Other surgical operations at the same time.
* Patients with pre-existing severe cardiac insufficiency, acute coronary syndromes, malignant hypertension and cardiogenic shock.
* Severe coagulation abnormality or severe anemia.
* Severe mental disorder.
* Malignant tumors.
* Pregnant or lactating.
* Increased risk of treatment for patients, according to investigators.
* Refuse to sign the informed consent form.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of MACCE | 3-month after the enrollment.
  MACCE includes all-cause of death, myocardial infarction, stroke and coronary revascularization surgery. The data will be obtained at 3-month follow-up, according to medical records of all patients.

SECONDARY OUTCOMES:
The incidence of all-cause of death | 3-month after the enrollment.
  The data will be obtained at 3-month follow-up, according to medical records of all patients.
The incidence of myocardial infarction | 3-month after the enrollment.
  The data will be obtained at 3-month follow-up, according to medical records of all patients.
The incidence of stroke | 3-month after the enrollment.
  The data will be obtained at 3-month follow-up, according to medical records of all patients.
The incidence of coronary revascularization surgery | 3-month after the enrollment.
  The data will be obtained at 3-month follow-up, according to medical records of all patients.
The length of postoperative ICU-stay | About 3 days after the operation.
  This outcome includes all days in ICU after the operation of all patients. The data will be recorded from the medical records.
The total length of stay in the hospital | About 7days after the operation.
  This outcome includes all days in the hospital of all patients. The data will be recorded from the medical records.
Changes of 6-min walk test results | 3-month after the enrollment.
  6-min walk test will be measured by stopwatches and metre rulers. The test assesses the overall response of all systems involved in exercise by measuring the distance the patient walks rapidly on a flat, hard surface over a period of six minutes.

OTHER OUTCOMES:
Total costs | 3-month after the enrollment.
  Total costs include CABG surgery, medications, examinations, management of complications during the first hospitalization and subsequent hospital admissions for cardiovascular problems. The data will be obtained from medical records and 3-month follow-up.
The incidence of adverse events | 3-month after the enrollment.
  Possible adverse events include ischemic pain, tissue damage (such as ulceration, gangrene), headache, bleeding events, neoplasm and accident (such as car accident, suicide) and etc. The data will be recorded from the medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yan, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiantong University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Yan Y, Zhao C, Niu J, Yan P, Li J, Wang D, Li G. Rationale and Design of the IMPROVE Trial: A Multicenter, Randomized, Controlled, Open-label, Blinded-endpoint Trial Assessing the Efficacy of Remote Ischemic Conditioning in Patients Undergoing Off-Pump Coronary Artery Bypass Grafting. Adv Ther. 2024 Jul;41(7):3003-3012. doi: 10.1007/s12325-024-02836-7. Epub 2024 Apr 15. PMID 38616242